CLINICAL TRIAL: NCT02877706
Title: French Registry of Adult Patients With Immune Thrombocytopenia and Autoimmune Hemolytic Anemia
Acronym: CARMEN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/12/0386
Record Dates: First submitted 2016-07-02; First posted 2016-08-24 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenia; Autoimmune Hemolytic Anemia
Keywords: Registry
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no specific intervention

SUMMARY:
CARMEN is a national, real-world clinical registry of all adult patients with incident diagnosis of Immune thrombocytopenia (ITP) or Autoimmune Hemolytic anemia (AIHA) patients in France. It is aimed at describing ITP and AIHA clinical features, assessing the real-world risk-benefit ratio of treatments and adherence to guidelines for ITP and AIHA management.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18+ year-old)
* newly diagnosed for ITP/AIHA or initiation of FOSFAMATINIB

Exclusion criteria:

- opposition to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric adult ITP and AIHA case recording in France, selected in centers of the French Referral Autoimmune Cytopenia Network. Both secondary and tertiary (referral) centers are participating (N=44).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-06; Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Immune thrombocytopenia (ITP) and AIHA | Baseline
  Number of new cases
Natural evolution and events | Baseline and follow-up
  Disease duration. Description of bleeding, infection, thrombosis events

SECONDARY OUTCOMES:
Response | 15 years
  platelet count >30 G/L and no bleeding
Complete rate | 15 years
  platelet count >30 G/L and no bleeding
Treatment lines | 15 years
  % of patients with each treatment by line of treatments
Adverse drug reactions | 15 years
  % of patients with adverse drug reaction reported by investigators
Bleeding | 15 years
  % of patients with bleeding during follow-up
Rescue treatment | 15 years
  % of patients with any treatment added during the exposure of ongoing treatment
Adherence to ITP management guidelines. | 15 years
  Percentage of patients who benefitted from the recommended examinations to detect secondary ITP and the percentage of patients who benefitted from the recommended first-line and second line treatments
Events | 15 years
  % of patients with other events of interest like cancer, death, infection, thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Moulis Guillaume, MD PhD, Principal Investigator — University Hopsital Toulouse
Locations (1):
- Service de Médecine Interne, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larue M, Moulis G, Rueter M, Audia S, Comont T, Terriou L, Viallard JF, Pan-Petesch B, Royer B, Bonnotte B, Galicier L, Lambotte O, Lefrere F, Cheze S, Ebbo M, Duong TA, Boutin E, Languille L, Mahevas M, Godeau B, Canoui-Poitrine F, Michel M. Efficacy and safety of dapsone in adult primary immune thrombocytopenia. Blood Adv. 2025 Apr 22;9(8):1976-1983. doi: 10.1182/bloodadvances.2024014939. PMID 39874521